CLINICAL TRIAL: NCT00937586
Title: Prostate Cancer Prospective Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Johns Hopkins University (Other); National Cancer Institute (NCI) (NIH); Wake Forest University (Other)
Responsible Party: Sponsor
Other Study IDs: HRPO#00-0327; R01CA112028 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Metastatic Prostate Cancer; Prostate Cancer Risk Assessment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, white cells, prostate tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly diagnosed patients: Patients with newly diagnosed prostate cancer.

SUMMARY:
The overall purpose of this research is to determine if certain genes increase the chance of developing prostate cancer and once diagnosed increase the chance of the prostate cancer spreading to other parts of the body.

DETAILED DESCRIPTION:
DNA will be isolated from each person and then studied for the presence of certain genes that may increase the chance of developing prostate cancer. Certain genes will also be studied in patients with known prostate cancer to determine if they increase the chance of cancer spreading to other parts of the body and decrease one's chance of being cured. Small differences in genes can slightly affect their ability to function. While these differences are normal, they may influence the way the cancer responds to therapy. An understanding of which genes increase (or decrease) the chance of being cured of a disease, such as prostate cancer, will improve our ability to take care of patients more effectively.

A second purpose of this study is to collect blood and cancer tissue for future studies. While the small differences in genes may be the best marker of bad cancer, it is also possible that proteins in blood or tumor may be a better marker.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients: 1. newly diagnosis of prostate cancer 2. untreated except for neoadjuvant systemic therapy.

Exclusion Criteria:

* Newly diagnosed patients: 1. inability to give informed consent

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed prostate cancer are being recruited for this study from Siteman Cancer Center radiation oncology, medical oncology and urology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1937 (Actual)
Dates: Start 2000-05; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Ability to recognize increased risk of metastatic prostate cancer based on specific genetic polymorphisms. | At the time of prostate cancer diagnosis

SECONDARY OUTCOMES:
Ability to predict risk for treatment failure based on analysis of specific polymorphisms. | At the time of prostate cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Drake, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States